CLINICAL TRIAL: NCT00192153
Title: A Randomized, Partially-Blinded, Placebo-Controlled Trial to Investigate Immune Responses Elicited by a Liquid Formulation of Influenza Virus Vaccine, (CAIV-T) in Healthy Adults 18 to 59 Years and Healthy Adults,60 Years/Older
Brief Title: Trial to Investigate Immune Responses Elicited by a Liquid Formulation of Influenza Virus Vaccine(CAIV-T)in Healthy Adults Aged 18 to 59 and Healthy Adults Aged 60 Years and Older
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D153 P003
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2006-10

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: CAIV-T or TIV

SUMMARY:
The purpose of this clinical study was to evaluate immune responses measuring antibodies in serum and secretions and cellular immune responses generated by CAIV-T vaccine in healthy adults aged 18 years and older as a means to develop assays for application in investigating potential immunological correlates of protection and/or establishing assays to measure vaccine take.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 59 years or > 60 years.
* Female subjects of childbearing potential who had a negative urine pregnancy test result prior to study vaccination. Females who were surgically sterile or post-menopausal did not require pregnancy testing.
* Adults who were determined by medical history, physical examination and clinical judgment eligible for this study. Subjects with stable pre-existing disease, defined as disease not requiring change in therapy or hospitalization within 12 weeks before receipt of study vaccination, will be eligible.
* Subjects who provided written informed consent after the nature of the study was explained.
* Subjects who were available for the duration of the study (from enrollment to study completion).
* Subjects who could be reached by study staff for the post-vaccination contact [via telephone, clinic or home visit].

Exclusion Criteria:

* For subjects > 60 years of age only:
* Subjects who resided in a nursing home or long-term care facility or other institution receiving skilled or semi-skilled nursing care. An ambulatory subject who resided in a retirement home or village was eligible for participation.
* Subjects with evidence of dementia or other severe cognitive impairment based on Mini Mental State Examination (MMSE) scores. Note: Prior to study vaccination, all subjects >60 years of age must have completed a MMSE.

For all study subjects:

* Subjects who were perceived to be unavailable or difficult to contact for evaluation of study visits during the study period.
* Subjects with a known or suspected disease of the immune system or those receiving immunosuppressive therapy, including systemic corticosteroids; or cytotoxic agents.
* Subjects who resided in the same household as an immunosuppressed or immunocompromised individual.
* Subjects with a documented history of hypersensitivity to egg or egg protein or any other component of the study vaccine, placebo or TIV.
* Subjects who had a current wheezing episode that was considered a change from the subject's usual clinical state.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240
Dates: Start 2001-07; Study Completion 2001-10

PRIMARY OUTCOMES:
To perform a variety of immunological assays using blood, serum, nasal washed an cells for application in the further investigation of immune responses generated by influenza virus vaccine, trivalent, types A and B, live, cold-adapted.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walker, MD, Principal Investigator — MedImmune LLC
Locations (2):
- United States (2):
  - West Coast Medical Associates, New Port Richey, Florida
  - University of VA Health Sciences Center, Charlottesville, Virginia